CLINICAL TRIAL: NCT02020577
Title: A Phase Ib Dose Escalation Study of Afatinib in Combination With Cetuximab in Patients With Advanced Solid Tumours
Brief Title: Trial of Afatinib (BIBW 2992) + Cetuximab in Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.122; 2012-005230-10 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-05

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Afatinib

ARMS (1):
- combination arm (Experimental): Patients to receive afatinib once daily plus weekly cetuximab infusion
  Interventions: Drug: Cetuximab( erbitux®); Drug: Afatinib

INTERVENTIONS:
Drug: Cetuximab( erbitux®) — once per week
Drug: Afatinib — once per day

SUMMARY:
The trial is divided in two parts, Part A and Part B. Part A will involve dose-finding of dose-limiting toxicity (DLT) and MTD in patients with advanced solid tumours. Part B will involve expansion of the MTD to 3 cohorts including non-small cell lung cancer squamous histology, recurrent/ metastatic squamous cell carcinoma of head and neck and other advanced solid tumours (except sarcomas).

ELIGIBILITY:
Inclusion criteria:

Part A only

1. Patients must have advanced malignant solid tumours that are metastatic or unresectable
2. At least one measurable or evaluable (non-measurable) lesion per RECIST 1.1 Part B only
3. Patients must have:

   1. measurable disease per RECIST 1.1
   2. diagnosis of one of the following

      * Advanced Non-Small Cell Lung Cancer -Squamous Histology (NSCLC-SQ) with no more than 2 lines of chemotherapy for advanced/metastatic disease ( prior EGFR directed treatment is permitted) or
      * Recurrent/Metastatic Squamous Cell Carcinoma of Head and Neck (R/M SCCHN) no more than 2 lines of chemotherapy for advanced disease and no more than 1 line of prior cetuximab permitted.

   or
   * Other malignant solid tumours except sarcomas (for metastatic colorectal cancer, only wild type KRAS are permitted) Part A and B
4. Age 18 years or older
5. Written informed consent that is consistent with ICH-GCP guidelines and local law.
6. Histological/Cytological confirmed diagnosis of malignant solid tumours (exclusion of sarcomas)
7. Advanced disease for whom standard treatment is ineffective or no longer effective
8. Recovered from previous therapy related AE to </= Grade 1 at the study entry (except, for stable sensory neuropathy </= Grade 2 and alopecia)
9. Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.
10. Adequate organ function as defined by the following criteria:

    * LVEF >50% or within institutional values
    * Absolute neutrophil count (ANC) >1500/ mm3
    * Platelet count >75.000/ mm3
    * Estimated creatinine clearance > 45ml/ min
    * Total bilirubin<1.5 times upper limit of institutional normal
    * Aspartate amino transferase (AST) or alanine amino transferase (ALT) <3 x upper limit of institutional normal (ULN) (if related to liver metastases< 5xULN)

Exclusion criteria:

1. Chemotherapy, biological therapy or investigational agents within 4 weeks prior to the start of study treatment.
2. Hormonal anti-cancer treatment within 2 weeks prior to the start of study treatment (continued use of anti-androgens and/or gonadorelin analogues [LHRH] is permitted)
3. Radiotherapy within 4 weeks prior to the start of study treatment, except as follows:

   1. Palliative radiation to target organs other than chest may be allowed up to 2 weeks prior to study treatment, and
   2. Single dose palliative treatment for symptomatic metastasis outside above allowance to be discussed with sponsor prior to enrolling.
4. Major surgery (as judged by the investigator) within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study
5. Known hypersensitivity to afatinib or the excipients of any of the trial drugs
6. History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of 3, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior start treatment.
7. Female patients of childbearing potential who:

   1. are nursing or
   2. are pregnant or
   3. are not using an acceptable method of birth control or do not plan to continue using this method throughout the study and/or do not agree to submit to pregnancy testing required by this protocol.
8. Any history of or concomitant condition that, in the opinion of the Investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug
9. Previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured.
10. Requiring treatment with any of the prohibited concomitant medications listed in the protocol that can not be stopped for the duration of trial participation
11. Known pre-existing interstitial lung disease
12. Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug (e.g. Crohn's disease, ulcerative colitis, chronic diarrhea, malabsorption)
13. Active hepatitis B infection (defined as presence of HepB sAg and/ or Hep B DNA), active hepatitis C infection (defined as presence of Hep C RNA) and/or known HIV carrier.
14. Prior participation in an afatinib clinical study, even if not assigned to afatinib treatment.
15. Meningeal carcinomatosis
16. Patients with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids or have been on stable dose of corticosteroids for at least 4 weeks before starting study treatment. Any symptoms attributed to brain metastases must be stable for at least 4 weeks before starting study treatment.
17. Any SPC listed contra-indications for cetuximab
18. Use of alcohol or drugs incompatible with patient participation in the study in the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- 1200.122.33001 Boehringer Ingelheim Investigational Site, Villejuif, France
- 1200.122.34001 Boehringer Ingelheim Investigational Site, Madrid, Spain

REFERENCES:
- [Derived] Gazzah A, Boni V, Soria JC, Calles A, Even C, Doger B, Mahjoubi L, Bahleda R, Ould-Kaci M, Esler A, Nazabadioko S, Calvo E. A phase 1b study of afatinib in combination with standard-dose cetuximab in patients with advanced solid tumours. Eur J Cancer. 2018 Nov;104:1-8. doi: 10.1016/j.ejca.2018.07.011. Epub 2018 Oct 1. PMID 30278378

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Uncontrolled, open label, 3+3 dose escalation (Part A) study of afatinib in combination with cetuximab, followed by an expansion phase in 3 cohorts of patients (Part B). Adverse Event (AE).
  CTCAE: Common Terminology Criteria for Adverse Events
Groups:
- Afatinib 30mg+Cetuximab 250 mg/m²: In each 21 day treatment cycle, patients were administered 30 mg Film-coated tablet daily afatinib in combination with cetuximab. An initial loading dose of cetuximab 400mg/m2 was administered intravenously at Day1 Cycle1, followed by cetuximab 250mg/m² weekly dose.
- Afatinib 40mg+Cetuximab 250 mg/m²: In each 21 day treatment cycle, patient were administered 40 mg Film-coated tablet daily afatinib in combination with cetuximab. An initial loading dose of cetuximab 400 mg/m2 was administered intravenously at Day1 Cycle1, followed by cetuximab 250mg/m² weekly dose.
Period: Overall Study
Arm/Group | Afatinib 30mg+Cetuximab 250 mg/m² | Afatinib 40mg+Cetuximab 250 mg/m²
Started | 3 | 55
Completed | 0 | 0
Not Completed | 3 | 55
Not completed — Progressive disease | 3 | 38
Not completed — Other AE or clinical progression | 0 | 15
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other than stated above | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set: This patient set includes all patients enrolled in the trial who were documented to have taken at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib 30mg+Cetuximab 250 mg/m² | Afatinib 40mg+Cetuximab 250 mg/m² | Total
Number analyzed (Participants) | 3 | 55 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (7.6) | 61.0 (11.4) | 61.1 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 20 | 20
  Male | 3 | 35 | 38

OUTCOME MEASURES:

1. Primary Outcome: MTD of Afatinib in Combination With Cetuximab Based on the Number of Patients With DLTs During the First Treatment Cycle (Afatinib).
Description: Maximum Tolerated Dose (MTD) of Afatinib in combination with cetuximab based on the number of patients with dose limiting toxicity (DLT) during the first treatment cycle (Dose escalation part). The MTD is defined as the highest dose level at which less than 33% of the patients experience DLT in first treatment cycle.
Time Frame: First 21 days treatment cycle
Population: Dose finding cohort treated set: This patient set includes all patients enrolled in part A of the trial who were documented to have taken at least one dose of study medication.
Measure: Number; unit: mg
Arm/Group | Afatinib 30mg+Cetuximab 250 mg/m² | Afatinib 40mg+Cetuximab 250 mg/m²
Number analyzed (Participants) | 3 | 6
mg | NA — MTD was not determined for this dose group. | 40

2. Primary Outcome: Dose Limiting Toxicities During Cycle 1
Description: Number of Patients With Dose Limiting Toxicity (DLT) Occurring during Cycle 1. The following drug related AEs qualified as DLT:
  1) CTCAE Grade ≥2 decrease in cardiac left ventricular function 2) CTCAE Grade 2 diarrhoea lasting for ≥7 days, despite appropriate use of standard antidiarrheal therapy based on Protocol Amendment 1 dated 22 Oct 2013 3) CTCAE Grade ≥3 diarrhoea despite appropriate use of standard anti-diarrheal therapy for at least 2 days. 4) CTCAE Grade ≥3 nausea and/or vomiting despite appropriate use of standard anti-emetics for at least 3 days 5) CTCAE Grade ≥3 rash despite standard medical management. 6) CTCAE Grade ≥3 fatigue lasting more than 7 days. 7) All other AEs of CTCAE Grade ≥3 (except alopecia and allergic reaction) that led to an interruption of afatinib and/or cetuximab dosing for more than 14 days until recovery to baseline or Grade 1, whichever was higher. 8) CTCAE Grade 4 hypomagnesemia or Grade 3 hypomagnesemia with clinically-significant sequelae
Time Frame: First 21-day treatment cycle
Population: Dose finding cohort treated set.
Measure: Number; unit: Participants
Arm/Group | Afatinib 30mg+Cetuximab 250 mg/m² | Afatinib 40mg+Cetuximab 250 mg/m²
Number analyzed (Participants) | 3 | 6
Participants | 0 | 0

3. Primary Outcome: MTD of Afatinib in Combination With Cetuximab Based on the Number of Patients With DLTs During the First Treatment Cycle (Cetuximab).
Description: Maximum Tolerated Dose (MTD) of Afatinib in combination with cetuximab based on the number of patients with DLTs during the first treatment cycle (Dose escalation part).
Time Frame: First treatment cycle
Population: Dose finding cohort treated set
Measure: Number; unit: mg/m2
Arm/Group | Afatinib 30mg+Cetuximab 250 mg/m² | Afatinib 40mg+Cetuximab 250 mg/m²
Number analyzed (Participants) | 3 | 6
mg/m2 | NA — MTD was not determined for this dose group. | 250

4. Secondary Outcome: Dose Limiting Toxicities During All Treatment Cycles
Description: Number of patients with DLT occuring during all treatment cycle is presented
Time Frame: All treatment cycle (each treatment cycle of 21 days)
Population: Treated Set
Measure: Number; unit: Participants
Groups:
- All Patients: Patients who were administered Afatinib 30mg+cetuximab 250 mg/m² plus the patients who were administered Afatinib 40mg+cetuximab 250 mg/m².
Arm/Group | Afatinib 30mg+Cetuximab 250 mg/m² | Afatinib 40mg+Cetuximab 250 mg/m² | All Patients
Number analyzed (Participants) | 3 | 55 | 58
Participants | 0 | 9 | 9

5. Secondary Outcome: Recommended Phase II Dose Based on the Number of Patients With Dose Limiting Toxicity Events (Cetuximab)
Description: MTD was deemed the recommended Phase II dose based on the number of patients with dose limiting toxicity events at all treatment cycles.
Time Frame: All treatment cycle (each treatment cycle of 21 days)
Population: Treated Set
Measure: Number; unit: mg/m2
Arm/Group | Afatinib 30mg+Cetuximab 250 mg/m² | Afatinib 40mg+Cetuximab 250 mg/m²
Number analyzed (Participants) | 3 | 55
mg/m2 | NA — MTD was not determined for this dose group. | 250

6. Secondary Outcome: Best Overall Response
Description: Best overall response (according to RECIST version 1.1) was defined as the best response recorded at any time from the first administration of afatinib or cetuximab to the End of Treatment (EOT).
  As Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI:
  Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; progression, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
Time Frame: Post baseline tumour-imaging was performed at every 6 weeks (in the week preceding the start of Cycles 3, 5, 7, 9, 11, etc.) until EOT; up to 19 months
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib 30mg+Cetuximab 250 mg/m² | Afatinib 40mg+Cetuximab 250 mg/m² | All Patients
Number analyzed (Participants) | 3 | 55 | 58
Percentage of participants
  Complete Response (CR) | 0.0 | 0.0 | 0.0
  Partial Response (PR) | 0.0 | 0.0 | 0.0
  Stable Disease (SD) | 66.7 | 52.7 | 53.4
  Progressive disease (PD) | 33.3 | 34.5 | 34.5
  Not evaluable (NE)/Missing | 0.0 | 12.7 | 12.1

7. Secondary Outcome: Objective Response
Description: Objective response was defined as the proportion of patients with measurable disease having at least a best overall response of complete response (CR) or partial response (PR), according to RECIST version 1.1.
  As Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI:
  Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; progression, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
Time Frame: as for outcome 6
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib 30mg+Cetuximab 250 mg/m² | Afatinib 40mg+Cetuximab 250 mg/m² | All Patients
Number analyzed (Participants) | 3 | 55 | 58
Percentage of participants | 0.0 | 0.0 | 0.0

8. Secondary Outcome: Disease Control Rate
Description: For patients with measurable disease, disease control was defined as the proportion of patients having at least a best overall response of CR, PR or stable disease (SD).
  As Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI:
  Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; progression, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression
Time Frame: as for outcome 6
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib 30mg+Cetuximab 250 mg/m² | Afatinib 40mg+Cetuximab 250 mg/m² | All Patients
Number analyzed (Participants) | 3 | 55 | 58
Percentage of participants | 66.7 | 52.7 | 53.4

9. Secondary Outcome: Recommended Phase II Dose Based on the Number of Patients With Dose Limiting Toxicity Events (Afatinib)
Description: as for outcome 5
Time Frame: All treatment cycle (each treatment cycle of 21 days)
Population: Treated Set
Measure: Number; unit: mg
Arm/Group | Afatinib 30mg+Cetuximab 250 mg/m² | Afatinib 40mg+Cetuximab 250 mg/m²
Number analyzed (Participants) | 3 | 55
mg | NA — MTD was not determined for this dose group. | 40

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after last drug administration, up to 19 months.
Arm/Group | Afatinib 30mg+Cetuximab 250 mg/m² | Afatinib 40mg+Cetuximab 250 mg/m² | All Patients
Serious Adverse Events (participants affected / at risk) | 1/3 | 31/55 | 32/58
Other Adverse Events (participants affected / at risk) | 3/3 | 54/55 | 57/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 30mg+Cetuximab 250 mg/m² (N=3) | Afatinib 40mg+Cetuximab 250 mg/m² (N=55) | All Patients (N=58)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Asthenia (General disorders) | 0 | 2 | 2
Mucosal inflammation (General disorders) | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 1
Bacterial infection (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1
Device related infection (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 2 | 2
Sepsis (Infections and infestations) | 0 | 3 | 3
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5 | 6
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Lymphoedema (Vascular disorders) | 0 | 2 | 2
Ophthalmoplegia (Eye disorders) | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 30mg+Cetuximab 250 mg/m² (N=3) | Afatinib 40mg+Cetuximab 250 mg/m² (N=55) | All Patients (N=58)
Anaemia (Blood and lymphatic system disorders) | 0 | 8 | 8
Lymphopenia (Blood and lymphatic system disorders) | 0 | 4 | 4
Tinnitus (Ear and labyrinth disorders) | 0 | 3 | 3
Dry eye (Eye disorders) | 0 | 5 | 5
Visual acuity reduced (Eye disorders) | 0 | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 3
Aphthous ulcer (Gastrointestinal disorders) | 0 | 3 | 3
Constipation (Gastrointestinal disorders) | 1 | 6 | 7
Diarrhoea (Gastrointestinal disorders) | 1 | 35 | 36
Dry mouth (Gastrointestinal disorders) | 0 | 8 | 8
Dysphagia (Gastrointestinal disorders) | 0 | 4 | 4
Nausea (Gastrointestinal disorders) | 0 | 10 | 10
Stomatitis (Gastrointestinal disorders) | 1 | 11 | 12
Vomiting (Gastrointestinal disorders) | 0 | 6 | 6
Asthenia (General disorders) | 0 | 17 | 17
Fatigue (General disorders) | 1 | 11 | 12
Mucosal inflammation (General disorders) | 0 | 9 | 9
Oedema peripheral (General disorders) | 0 | 5 | 5
Pain (General disorders) | 0 | 4 | 4
Pyrexia (General disorders) | 0 | 12 | 12
Xerosis (General disorders) | 0 | 3 | 3
Hepatocellular injury (Hepatobiliary disorders) | 0 | 5 | 5
Conjunctivitis (Infections and infestations) | 1 | 5 | 6
Folliculitis (Infections and infestations) | 0 | 18 | 18
Paronychia (Infections and infestations) | 1 | 17 | 18
Urinary tract infection (Infections and infestations) | 0 | 3 | 3
Blood phosphorus decreased (Investigations) | 0 | 4 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 17 | 17
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 10 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 26 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4
Dizziness (Nervous system disorders) | 0 | 4 | 4
Headache (Nervous system disorders) | 1 | 2 | 3
Anxiety (Psychiatric disorders) | 0 | 3 | 3
Depression (Psychiatric disorders) | 0 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 9 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 7
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 22 | 24
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 14 | 16
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 5 | 6
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 11 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 11 | 12
Rash (Skin and subcutaneous tissue disorders) | 1 | 7 | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 7 | 7
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 14 | 14
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 10 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.